CLINICAL TRIAL: NCT06362694
Title: Study of the Rechallenge Concept in Patients With BRAF-positive Anaplastic Thyroid Cancer After Progression on Anti-BRAF Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Ernest Dzhelialov, Oncologist, Saint Petersburg State University, Russia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 34
Record Dates: First submitted 2024-03-28; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Anaplastic Thyroid Cancer
Keywords: anaplastic thyroid cancer; rechallenge; dabrafenib; trametinib; targeted therapy
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic | interventions — dabrafenib; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Patients with BRAF-positive anaplastic thyroid cancer who were previously treated with dabrafenib and trametinib (with a clinical or objective response at the start of treatment) and later with tumor progression during anti-BRAF therapy with the transition to at least one line of chemotherapy (treatment with taxane-containing regimens is mandatory) followed by progression on it.
  Interventions: Drug: Dabrafenib + Trametinib

INTERVENTIONS:
Drug: Dabrafenib + Trametinib — Dabrafenib is an inhibitor of some mutated forms of BRAF kinases. Trametinib is a reversible inhibitor of mitogen-activated extracellular signal-regulated kinase 1 (MEK1) and MEK2 activation and of MEK1 and MEK2 kinase activity. Dabrafenib and trametinib target two different kinases in the RAS/RAF/MEK/ERK pathway. Use of dabrafenib 623 and trametinib in combination resulted in greater growth inhibition of BRAF V600 mutation-positive tumors.

SUMMARY:
This pilot phase 2 study evaluates the effectiveness and safety of the Rechallenge concept in patients with BRAF-positive anaplastic thyroid cancer after progression on anti-BRAF therapy. Patients with BRAF-positive anaplastic thyroid cancer who were previously treated with dabrafenib and trametinib (with a clinical or objective response at the start of treatment) and later with tumor progression during anti-BRAF therapy and subsequent lines of chemotherapy are scheduled to undergo targeted therapy (repeated administration of dabrafenib and trametinib in standard doses) and evaluate the outcomes according to the primary and secondary endpoints.

DETAILED DESCRIPTION:
The aim of the study was to demonstrate the efficacy and safety of the rechallenge concept in patients with BRAF-positive anaplastic thyroid cancer after progression on anti-BRAF therapy.

Scientific hypothesis: rechallenge in patients with BRAF-positive anaplastic thyroid cancer after progression on anti-BRAF therapy is effective and safe.

Trial design, materials and methods: this study is a pilot phase 2 study. This study is prospective and open-label.

Patients with BRAF-positive anaplastic thyroid cancer who were previously treated with dabrafenib and trametinib (with a clinical or objective response at the start of treatment) and later with tumor progression during anti-BRAF treatment with the transition to at least one line of chemotherapy (treatment with taxane-containing regimens is mandatory) followed by progression on it. Patients who meet the criteria and with no initial resistance to anti-BRAF therapy are scheduled to undergo targeted therapy (repeated administration of dabrafenib and trametinib in standard doses) and evaluate outcomes according to primary and secondary endpoints.

The control will be carried out by monitoring the initial state in dynamics. Before starting investigational therapy, data will be recorded for each patient in an individual registration card.

Before starting investigational therapy, clinical and laboratory parameters will be evaluated and computed tomography of the brain, neck, thoracic and abdominal cavities with intravenous contrast (baseline) will be performed.

Mutations in the BRAF V600 gene, microsatellite instability (MSI) and PD-L1 expression will be determined in the tumor material (first of all), and the following molecular genetic variants will be determined in the second place (planned): RET, NTRK, ALK, ROS1.

Investigational therapy includes dabrafenib 150 mg 2 times a day daily, trametinib 2 mg 1 time a day daily.

Duration of treatment: until progression or intolerable toxicity.

Follow-up period of patients:

* duration of the initial follow-up period: taking drugs for 10 days, followed by an assessment of the effect using tumor imaging methods;
* follow-up during active treatment in the framework of the study with tumor reduction after day 10 - continuation of targeted therapy until progression or intolerable toxicity;
* patient survival monitoring - documenting subsequent lines of antitumor treatment before the patient's death or loss of contact with him;
* patient safety monitoring is the period of research therapy, 30 and 90 days from the date of the final dose (provided there is no next line of antitumor treatment, during the next line, safety monitoring is discontinued).

Assessment of the response to treatment (assessment of clinical and laboratory parameters, computed tomography of the brain, neck, chest and abdominal cavity with intravenous contrast) will be carried out after 10 days, then - according to the decision of the research team. Based on the results of the control study, the response to treatment will be evaluated according to the RECIST 1.1 criteria. Patients who meet the criteria for progression will be excluded from the study.

When converting a tumor to resectability and planning surgical treatment, it is recommended to suspend taking the drug trametinib 5 days before surgery and resume taking it 3-5 days after. There is no correlation between dabrafenib and complications associated with surgical treatment, and no interruptions in treatment are required.

ELIGIBILITY:
Inclusion Criteria:

* immunohistochemically verified anaplastic thyroid cancer;
* presence of a mutation in the BRAF V600 gene;
* documented progression during targeted therapy with dabrafenib + trametinib;
* documented progression during at least one line of chemotherapy (use of taxane-containing chemotherapy is mandatory);
* age ≥ 18 years;
* ECOG performance status 0-2;
* adequate function of internal organs and bone marrow;
* ability to give written informed consent.

Exclusion Criteria:

* primary resistance (absence of initial clinical and radiological response to therapy with dabrafenib and trametinib (response criteria - primary objective response according to RECIST 1.1 criteria and duration of response of at least 3 months);
* absence of taxane-containing chemotherapy as second or third line;
* contraindication to taking any of the study drugs (including severe toxicity that occurred during a previous dose, which led to discontinuation of treatment);
* patients with unsatisfactory functional status (ECOG 3-4);
* pregnancy and breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 10 days, then each month from date of treatment initiation until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months
  The proportion of participants with a partial or complete response to the therapy. It is determined according to the RECIST criteria.
Progression-Free Survival | 6-month, 1-year, 2-year
  The time from the date of initiation of treatment to the radiological progression or death of the patient for any reason.
Safety and Tolerability assessment (Incidence of Treatment-Emergent Adverse Events) | Each visit (every 21 days) assessed up to 48 months
  Safety assessment will be assessed on the basis of adverse events (according to CTCAE 5.0)

SECONDARY OUTCOMES:
Overall survival | 6-month, 1-year, 2-year
  The time from the start date of treatment to the death of the patient for any reason.
The assessment of conversion to resectability | Each month from date of treatment initiation until the date of first documented progression or date of death from any cause, whichever came first , assessed up to 48 months
  The proportion of participants with an initially unresectable or potentially resectable tumor who have moved to a resectable during treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Petersburg State University Hospital, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code